CLINICAL TRIAL: NCT00188903
Title: Diastolic Dysfunction and Atrial Fibrillation in Patients Undergoing Coronary Revascularization Surgery
Brief Title: Diastolic Dysfunction and Atrial Fibrillation in CABG Surgery
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: George Djaiani, Toronto General Hospital, University Health Network
Other Study IDs: UHN REB 03-0873-A
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2010-08-05 (Estimated); Status verified 2008-04

CONDITIONS: Heart Disease; Atrial Fibrillation
Keywords: Cardiac Surgery; Diastolic Dysfunction; Atrial Fibrillation
MeSH Terms: conditions — Heart Diseases; Atrial Fibrillation

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: Diastolic measurements during TEE — Transesophageal echocardiography with diastolic measurements

SUMMARY:
Left ventricular (LV) diastolic dysfunction is a common manifestation of heart disease that is responsible for significant morbidity and mortality.It is present when the ventricular filling is impaired as a result of delayed relaxation or decreased compliance. During Coronary artery bypass grafting (CABG) surgery, LV diastolic dysfunction is a frequent occurrence. Failure of the left ventricle to dilate normally causes an increase in LV filling pressure. Atrial fibrillation (AF) is a common complication after cardiac surgery affecting 20-30% of patients undergoing coronary revascularization procedures. AF is associated with significant morbidity and mortality and has been identified as a causative factor of increased length of both hospital and intensive care unit (ICU) stay after CABG surgery, resulting in increased resource utilization and medical care costs.The primary aim of this study is to determine if patients with preoperative diastolic dysfunction are exposed to higher risk of AF after coronary revascularization surgery.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for elective CABG or OPCAB surgery
* signed informed consent

Exclusion Criteria:

* Patients with a history of previous heart surgery and/or undergoing valvular heart surgery.
* Patients with preoperative atrial fibrillation.
* Patients in whom TEE is contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elective coronary artery bypass graft patients either on or off pump in acute care centre
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2004-03; Primary Completion 2007-11 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Is to determine if patients with preoperative diastolic dysfunction are exposed to higher risk of AF after coronary revascularization surgery. | pre and post operative

SECONDARY OUTCOMES:
Is to determine if diastolic dysfunction and AF are associated with increased perioperative cardiac morbidity and reduced event-free survival. | post operative until discharge

CONTACTS AND LOCATIONS:
Overall Officials: George N Djaiani, MD, Principal Investigator — Toronto General Hospital, Univsersity Health Network
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Ashes CM, Yu M, Meineri M, Katznelson R, Carroll J, Rao V, Djaiani G. Diastolic dysfunction, cardiopulmonary bypass, and atrial fibrillation after coronary artery bypass graft surgery. Br J Anaesth. 2014 Nov;113(5):815-21. doi: 10.1093/bja/aeu208. Epub 2014 Jul 8. PMID 25005721